CLINICAL TRIAL: NCT06742242
Title: The Use of Non-Indocyanine Green-Enhanced Lymphatic Vessels for Supermicrosurgical Lymphaticovenous Anastomosis: a Propensity-Score-Matched Outcome Analysis
Brief Title: The Use of Non-ICG-Enhanced Lymphatic Vessels for LVA
Acronym: ICG LVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202400198B0
Record Dates: First submitted 2024-10-04; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-04

CONDITIONS: Lymphedema
Keywords: propensity score matching; LVA; Supermicrosurgery; lymphaticovenous anastomosis; lymphovenous bypass
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The Use of Non-ICG-Enhanced Lymphatic Vessels for LVA (Experimental): The use of non-ICG-enhanced lymphatic vessels for LVA
  Interventions: Procedure: lymphaticovenous anastomosis

INTERVENTIONS:
Procedure: lymphaticovenous anastomosis — supermicrosurgical lymphatic vessel to recipient ven lumen-to-lumen coaptation

SUMMARY:
The aim of the present study was to investigate the impact of non-ICG(+) LVs on the outcomes after LVA compared to ICG(+) LVs with propensity-score-match analysis.

DETAILED DESCRIPTION:
It is a common belief among lymphatic supermicrosurgeons that LVA should only be performed with indocyanine green-enhanced (ICG(+)) LVs since such LVs are considered functional and are suitable for achieving better outcomes. However, in moderate to advance lymphedema patients, the use of non-ICG(+) LVs are inevitable despite efforts to identified ICG(+) LVs with ICG lymphography10, magnetic resonance (MR) lymphangiography11, or ultrasound12. In a previous study, it was suggested that a non-ICG(+) but flow-positive LV should also be considered functional because the functionality of an LV should be determined by its capability to transport lymph instead of ICG(+) lymph. Therefore, non- ICG(+) but flow-positive LVs should also be used for LVA to maximize the outcome13. This hypothesis was further supported by a recent article emphasizing the concept of a lymphatic-based lymphosome14, where it has been demonstrated that a functional LV will not become ICG(+) when ICG is not injected in the region being drained by this particular LV. It offers an explanation as to why a supposedly functional LV is not enhanced by ICG.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lymphatic-related diseases at Kaohsiung Chang Gung Memorial Hospital from September 2015 to March 2023.
* Patients who underwent LVA for unilateral lower-limb lymphedema.

Exclusion Criteria:

* Primary lymphedema
* Bilateral lower limb lymphedema
* History of previous treatment for lymphedema (LVA, vascularized lymph node transfer (VLNT), liposuction, or excisional therapy such as the Charles procedure) - Those that were lost to follow-up.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Volume change after LVA. | 6/12 months
  The primary endpoint was the volume change at 6/12 months after LVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No